CLINICAL TRIAL: NCT04289493
Title: DUbbing Language-therapy CINEma-based in Aphasia Post-Stroke (DULCINEA). A Feasibility Cross-over Pilot-trial
Brief Title: DUbbing Language-therapy CINEma-based in Aphasia Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Pontificia Comillas (Other); Asociación Afasia Activa (Other); La Caixa Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DULCINEA
Record Dates: First submitted 2020-02-20; First posted 2020-02-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Aphasia, Post-Ictal
Keywords: Rehabilitation; Word dubbing; Functional communication
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Two groups with 27 patients in each one. Group 1 starts therapy in the first 3 months since study inclusion and from months 3-6 is group 2 control. Group 2 starts language therapy from months 3-6, serving previously as group 1 control.
Who Masked: Outcomes Assessor
Masking Description: A psychologist blinded to the patient´s clinical characteristics and study groups performs the outcome questionnaires three times for each patient during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: first to receive therapy (Experimental): 27 patients that will receive study specific speech therapy in the first 3 months since study inclusion. From months 3-6 they will be group 2 controls.
  Interventions: Other: Language and functional communication therapy
- Group 2: second to receive therapy (Experimental): 27 patients that will receive study specific speech therapy during months 3-6 since study inclusion. During the first 3 months of the study period, they will be group 1 controls.
  Interventions: Other: Language and functional communication therapy

INTERVENTIONS:
Other: Language and functional communication therapy — 17 therapy sessions in which the patients will be asked to dubb words or sentences from television series previously considered functionally meaningful for them.

SUMMARY:
The DULCINEA study aims to develop and validate a new therapy that integrates essential language characteristics and functional communication by dubbing scenes from television series that represent daily situations. It will be a randomized, crossed over, interventional pilot study recruiting 54 patients with poststroke nonfluent aphasia. Patients will be treated individually in 40-minute sessions twice a week for 8 weeks. In each session, a speech therapist and an actor will select the clips with muted words or sentences that have been detected as functionally meaningful for each patient. Outcomes will be assessed as significant differences in two aphasia tests.

DETAILED DESCRIPTION:
The DULCINEA study aims to develop and validate a new therapy that integrates essential language characteristics and functional communication by dubbing scenes from TV series that represent daily situations. It will be a randomized, crossed over, interventional pilot study recruiting 54 patients with poststroke nonfluent aphasia from the departments of Neurology and Rehabilitation from La Paz University Hospital and also from the "Afasia Activa" association. After meeting all inclusion and none of the exclusion criteria and signing informed consent, patients will be randomised (1:1) in two different treatment groups. The first group will receive therapy within the first 3 months of their inclusion with a subsequent period of another 3 months without therapy (thus, serving as group 2 controls). Group 2 will initiate therapy after 3 months since their inclusion (serving as group 1 controls during the first 3 months). Therapy consists of 17 sessions performed in a eight week period (1 baseline session and 16 dubbing sessions), each lasting 40 minutes, in which the patient will be asked to dubb words or sentences previously selected and considered as functionally meaningful for them. These words will be chosen through an online survey performed by a representative group of aphasic patients and the study patients´own relatives in the baseline treatment session. Outcomes will be assessed as significant differences in two aphasia tests (CAL questionnaire and the BDAE).

ELIGIBILITY:
Inclusion Criteria:

* nonfluent aphasia due to unilateral stroke in the left hemisphere without neuroimaging evidence of lesions in the right hemisphere.
* the patient should have received a standard program of conventional speech therapy after stroke, remaining with aphasia with the following characteristics: severely restricted language, poor repetition (even for single words), not exceeding the 70th percentile in the Boston Diagnostic Aphasia Examination (BDAE) for repetition. Moderately preserved language comprehension: listening comprehension exceeding the 15th percentile of BDAE (average score obtained in three areas: word comprehension, commands and complex ideational material).
* Signed informed consent.

Exclusion Criteria:

* Any clinical condition (short life expectancy, coexisting disease) or other characteristics that precluded appropriate follow-up.
* Participation in any therapeutic trial evaluating poststroke recovery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Communicative Activity Log (CAL) questionnaire | Changes in score at six months
  Questionnaire that evaluates quantity and quality of aphasic patient communication, with 18 different questions in each item. Each question belonging to these two items is answered as a 6 point scale, where 0 is the worst and 5 is the best score.
Boston Diagnostic Aphasia Examination (BDAE) | Changes in score at six months
  Neuropsycological battery that evaluates language skills based on perceptual modalities (auditory, visual, and gestural), processing functions (comprehension, analysis, problem-solving), and response modalities (writing, articulation, and manipulation). There are five subtests which include: conversational and expository speech, auditory comprehension, oral expression, reading, and writing. Its results can be used to classify patient's language profiles into one of the localization based classifications of aphasia, and it also provides a severity rating.

SECONDARY OUTCOMES:
General Health Questionnaire (GQH-12) | Changes in score at six months
  The General Health Questionnaire (GHQ) is a psychometric screening tool to identify common psychiatric conditions. It comprises 12 questions, each one with a four point scale answer.
Stroke and aphasia Quality of Life Scale (SAQOL-39) | Changes in score at six months
  SAQOL-39 is an interview-administered self-report scale that comprises the 49 items of the SS-QOL (modified to be communicatively accessible to people with aphasia) and 4 additional items that measure speech comprehension, difficulties with decision-making and and impact of language problems on family and social life. Questions are answered with a five point scale.
Western Aphasia Battery Revised (WAB-R) | Changes in score at six months
  This neuropsycological test assesses linguistic and non-linguistic skills comprised of 8 subtest (32 short tasks). It identifies aphasia and classifies the type and severity of aphasia disorders.
Stroke Aphasic Depression Questionnaire (SADQ10) | Changes in score at six months
  This is a brief questionnaire with 10 items testing depression symptoms within the last week in aphasic patients. Each item scores in a four point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuentes B, de la Fuente-Gomez L, Sempere-Iborra C, Delgado-Fernandez C, Tarifa-Rodriguez A, Alonso de Lecinana M, de Celis-Ruiz E, Gutierrez-Zuniga R, Lopez-Tappero J, Martin Alonso M, Pastor-Yborra S, Rigual R, Ruiz-Ares G, Rodriguez-Pardo J, Virues-Ortega J, Borobia AM, Blanco P, Bueno-Guerra N. DUbbing Language-therapy CINEma-based in Aphasia post-Stroke (DULCINEA): study protocol for a randomized crossover pilot trial. Trials. 2022 Jan 6;23(1):21. doi: 10.1186/s13063-021-05956-5. PMID 34991688